CLINICAL TRIAL: NCT06513676
Title: The First Affiliated Hospital of Xinjiang Medical University
Brief Title: Super Selective Adrenal Artery Embolization for Primary Aldosteronism: a Prospective Cohort Study(SAAE-PA)
Status: Recruiting | Type: Observational
Sponsor: Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Xiang Xie, Xiangxie, MD,Professor, The First Affiliated Hospital Of XinJiang Medicial University, Xinjiang Medical University
Other Study IDs: 240528-09
Record Dates: First submitted 2024-06-12; First posted 2024-07-22 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-06

CONDITIONS: Primary Aldosteronism; Super Selective Adrenal Arterial Embolization
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Super selective adrenal artery embolization: SAAE for primary aldosteronism
- adrenectomy: Surgery to remove part of the adrenal gland
- Standard drug therapy: Drug treatment of primary aldosteronism

SUMMARY:
The objective of this study was to evaluate the efficacy and safety of adrenal vein blood extraction for primary aldosteronism classification and adrenal artery embolization in the treatment of primary aldosteronism, to provide new evidence plan for the diagnosis and treatment of primary aldosteronism, and to promote the development of adrenal artery embolization as a new treatment for primary aldosteronism.

DETAILED DESCRIPTION:
As one of the causes of refractory secondary hypertension, primary aldosteronism is usually treated with drug therapy and adrenalectomy, but the therapeutic effect of these regimens is limited in some people. Adrenal vein blood collection is a method to identify the types of primary hyperaldosteronism by comparing the ratio of aldosterone in venous blood by selective catheterization into adrenal vein. Superselective adrenal artery embolization is a catheter-based percutaneous cavitary procedure in which ethanol is selectively injected into the adrenal artery to ablate part of the adrenal gland. Recently, it has been used as an alternative therapy for patients with unilateral aldosterone-producing adenomas as well as idiopathic hyperaldosteronism without obvious adenomas. This is a prospective, multicenter, randomized controlled study in Xinjiang to explore the potential of SAAE as a treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years old;
* Primary hyperaldosteronism was diagnosed in strict accordance with the 2016 International Endocrine Society clinical guidelines;
* Refusal of medication due to adverse reactions, refusal of adrenal resection due to surgical risk, or persistent hyperaldosteronism and cortical insufficiency after adrenal resection;
* The patients and their families were introduced in detail to all the current treatment methods for primary aldosteronism, and the adrenal artery embolization was voluntarily accepted;

Exclusion Criteria:

* A history of severe hypersensitivity to contrast media;
* There are serious complications of liver disease, such as thrombocytopenia, esophageal variceal bleeding, etc;
* Renal insufficiency (serum creatinine > 176mmol/L or estimated glomerular filtration rate < min.1.73m2);
* Combined with other secondary hypertension, such as pheochromocytoma, hypercortisolism, renal vascular hypertension (such as renal artery stenosis), renin secretory tumor, renal parenchymatous hypertension, drug-induced hypertension (such as long-term use of glucocorticoids, contraceptives, estrogens, herbs containing glycyrrhizin), pregnancy hypertension and other secondary hypertension;
* Hereditary diseases: such as false aldosteronism (Liddle syndrome), Bartter syndrome, familial hypokalemia and hypomagnesemia (Gitelman syndrome);
* Cerebral apoplexy, myocardial infarction and stent implantation occurred in the past 3 months;
* Serious other basic, such as heart dysfunction (grade IV), acute infection, autoimmune diseases, various malignant tumors and so on;
* Participated in other clinical trials within the past 3 months;
* Individual pregnancy, nursing or planning pregnancy;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Hypertensive patients were willing to participate and then hospitalized for further evaluation. Antihypertensive medications that affect the renin-angiotensin-aldosterone system were stopped for two weeks, diuretics and MRA were withdrawn for at least 4 weeks before ARR testing. Hypertensive patients were prescribed with verapamil and/or terazosin based on Endocrine Society Clinical Practice Guideline. Patients with positive aldosterone-to-renin ratio underwent one of the following confirmatory tests: saline infusion test or captopril inhibition test. Adrenal CT scan and adrenal venous sampling (AVS) were performed for subtype classification of the PA. The PA patients were counseled on the various treatment options, including surgery, medications, and adrenal artery ablation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Complete biochemical cure of PA | 6 months post intervention
  Complete biochemical cure of PA, defined (whilst off medications that might alter serum potassium or the RAS) by both:
  1. Normalisation of serum potassium, and
  2. Normalisation of ARR, or
  3. Elevated ARR and i). Baseline PAC <190pmol/L, or ii). Normal confirmatory test (as defined in the inclusion criteria)
Complete clinical cure of PA | 6 months post intervention
  Complete clinical cure of PA, defined as normotension without antihypertensive medication
  These criteria have been defined in the international consensus PASO statement8, which has become the established yardstick by which PA cure is judged. In this, normotension is defined, in accordance with the European Society of Hypertension guidelines22, as <140/80 in the office, <135/85 at home or daytime ambulatory monitoring and <130/80 for 24h ambulatory blood pressure monitoring (24hABPM).

SECONDARY OUTCOMES:
Changes in ambulatory blood pressure and baseline blood pressure | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  24-hour ambulatory blood pressure and office systolic and diastolic pressure
Change of the number of antihypertensive medications | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  Difference in the change of the number of antihypertensive medications
Adverse events | Reported throughout the study period. Approximately 2 years
  Will be directly sought at each study visit through history and physical examination where appropriate Subjects will be encouraged to report between study visits and will have a mechanism to do so Will be classified by system, seriousness, causal relationship and expectedness according to the Common Terminology Criteria for Adverse Events v5.0 (CTCAE)
Readmission rate | Reported throughout the study period. Approximately 2 years
  Readmission rate, defined as readmission for primary aldosteronism
Change of blood electrolytes (K+, Na +) | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  Difference in the change of blood electrolytes (K+, Na + in mmol/L)
Change of plasma aldosterone | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  Difference in the change of plasma aldosterone (pg/mL)
Change of plasma cortisol | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  Difference in the change of plasma cortisol (nmol/L)
Change of plasma renin measured | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  Difference in the change of plasma renin (pg/ml)
Change of liver enzymes | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  Difference in the change of liver enzymes (ALT, AST in IU/L)
Change of kidney function | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  Difference in the change of serum creatinine in umol/L
Change of fasting blood glucose | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  Difference in the change of fasting blood glucose in mmol/L
Change of lipids profiles | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  Difference in the change of lipids profiles (TC, HDL-C, LDL-C, TG) in mmol/L
Change of 24-h urine microalbumin | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  Difference in the change of 24-h urine microalbumin (mg/L)
Change of 24-h 24-h urine creatinine | 1 day, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months
  Difference in the change of 24-h urine creatinine (umol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang, China